CLINICAL TRIAL: NCT05780190
Title: Clinical Observation of New Artificial Liver CABA System (BS330+CA280) in the Treatment of End-stage Liver Disease With Inflammation
Brief Title: Clinical Observation of CABA System in the Treatment of End-stage Liver Disease With Inflammation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CABA STUDY
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: To Evaluate the Clinical Efficacy and Safety of the New ALSS

STUDY DESIGN:
Intervention Model Description: CABA+PE+standard drug therapy and PP+PE+standard drug therapy
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABA group (Experimental): new artificial liver CABA system (BS330+CA280) combined with plasma exchange
  Interventions: Device: New artificial liver CABA system (BS330+CA280) +PE
- control group (Experimental): BS330 combined with plasma exchange
  Interventions: Device: New artificial liver CABA system (BS330+CA280) +PE

INTERVENTIONS:
Device: New artificial liver CABA system (BS330+CA280) +PE — The new artificial liver CABA system (BS330+CA280) combioned plasma exchange in the treatment of end-stage liver disease with inflammatory status
  Other Names: standard drug therapy

SUMMARY:
End-stage liver disease (ESLD) refers to the late stage of liver disease caused by various chronic liver damage. ESLD is an important cause of global incidence rate and mortality, which has a significant impact on the health care system.

ESLD is associated with various types of immune dysfunction. The artificial liver support system (ALSS) is an extracorporeal support system that temporarily and partially replaces the partial function of the liver. Its treatment mechanism is to remove all kinds of harmful substances, supplement essential substances, improve the internal environment, create conditions for hepatocyte regeneration and liver function recovery, or use it as a symptomatic support treatment method during the perioperative period of liver transplantation. In this study, we plan to use BS330 for plasma bilirubin adsorption. On this basis, we will add a CA280 cytokine adsorption column to establish a new artificial liver combination model CABA for the immune inflammatory damage mechanism of liver failure.

DETAILED DESCRIPTION:
End-stage liver disease (ESLD) refers to the late stage of liver disease caused by various chronic liver damage. Its main feature is that the liver function cannot meet the physiological needs of the human body. Its scope includes the end stage of various chronic liver diseases, including chronic plus acute liver failure (ACLF), acute decompensation of cirrhosis (ADC), chronic liver failure (CLF) and hepatocellular carcinoma. ESLD is an important cause of global incidence rate and mortality, which has a significant impact on the health care system.

ESLD is associated with various types of immune dysfunction. The symptoms of these immune dysfunction are called cirrhosis-related immune dysfunction (CAID), characterized by immune deficiency and systemic inflammation caused by the continuous and inappropriate activation of immune cells. In compensated cirrhosis, even without intestinal bacterial translocation, the damage-related molecular patterns (DAMPs) released by necrotic hepatocytes can activate the immune system and cause systemic inflammation. During the decompensation period, the bacterial products produced by intestinal bacterial translocation enhance immune activation and increase the expression of pro-inflammatory cytokines and immune cell activation antigens in the circulation. Cytokines are the key components of the immune system, with a variety of characteristics and biological functions. Systemic inflammation associated with CAID is associated with increased circulating levels of pro-inflammatory cytokines such as interleukin (IL) - 6. Studies have shown that there is a relationship between the severity of immune disorders and the prognosis of liver cirrhosis. The levels of IL-6, IL-10 and IL-17 are increased in liver cirrhosis.

The artificial liver support system (ALSS) is an extracorporeal support system that temporarily and partially replaces the partial function of the liver. Its treatment mechanism is to remove all kinds of harmful substances, supplement essential substances, improve the internal environment, create conditions for hepatocyte regeneration and liver function recovery, or use it as a symptomatic support treatment method during the perioperative period of liver transplantation. Plasma bilirubin adsorption is the specific adsorption of bilirubin through anion resin adsorption column, which can effectively reduce the level of bilirubin and bile acid, thus improving the internal environment of the machine and helping the further repair of damaged liver cells. Cytokine adsorption is designed to reduce the level of cytokines represented by IL-6 through the cytokine adsorption column. In clinical practice, it is mainly used to reduce the level of circulating pro-inflammatory cytokines and early harmful effects in the first few hours and days of treatment of infectious shock, so as to improve the treatment effect of patients. In this study, we plan to use BS330 for plasma bilirubin adsorption. On this basis, we will add a CA280 cytokine adsorption column to establish a new artificial liver combination model CABA for the immune inflammatory damage mechanism of liver failure. This treatment model can not only absorb bilirubin, but also effectively remove more inflammatory factors. In this study, patients with end-stage liver disease and inflammatory status will be selected as the observation object, and the new CABA combination will be used for treatment, and the clinical effectiveness and safety of this treatment mode will be evaluated, aiming to provide evidence-based medical evidence for the clinical application and promotion of this treatment mode.

ELIGIBILITY:
Inclusion Criteria:

① Age 18-70;

② Patients with end-stage liver disease, including patients with acute decompensation of cirrhosis, chronic liver failure and patients with chronic and acute liver failure in Child-Pugh grade B-C;

A. Acute decompensation of liver cirrhosis:

1. ALB<35 g/L; A / G <1.0;
2. TBIL> 120 μ mol / L;
3. ALT> 1 × ULN and/or AST>1 × ULN;
4. PTA <60%
5. Ascites or hepatic encephalopathy or bleeding from esophageal varices;

B. Chronic liver failure:

1. The basis of chronic liver disease: decompensated cirrhosis;
2. Time of onset: unlimited;
3. Hepatic encephalopathy: with or without;
4. Coagulation: PTA ≤ 40% or INR ≥ 1.5;
5. Jaundice>171.1umol/L;

C. Chronic plus acute liver failure:

1. Chronic liver disease is based on: chronic hepatitis or decompensated cirrhosis;
2. Time of onset:<4 weeks;
3. Hepatic encephalopathy: with or without;
4. Coagulation: PTA ≤ 40% or INR ≥ 1.5;
5. Jaundice: TBIL ≥ 171 μ Mol/L or daily increase ≥ 17.1 μ mol/L

   ③ Inflammation status: the following 4 items meet any 2 items
   1. PCT≥0.50 μ g/L
   2. CRP≥40 mg/L
   3. IL-6 > 5 × ULN
   4. IL-8 > 5 × ULN

      ④ Understand and voluntarily sign the informed consent form approved by the Ethics Committee.

      Exclusion Criteria:
      * Patients with liver malignant tumor and other tumors;

        * People with HIV infection or other immunodeficiency diseases;

          * Pregnant or lactating women;

            * Patients with autoimmune disease, unstable stage of infarction caused by cardio-cerebrovascular accident, history of organ transplantation and other organ dysfunction or failure; ⑤ Patients with other serious complications (such as active bleeding, diffuse intravascular coagulation); ⑥ Those who are unable to return to the hospital for further consultation and follow-up regularly according to the research plan;

              * Those who fail to comply with the research arrangement and sign the informed consent form; ⑧ Other conditions judged by the researcher not suitable for the group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-03-08 (Estimated); Study Completion 2024-03-08 (Estimated)

PRIMARY OUTCOMES:
non-transplantation mortality | 1 year
  the 28-day and 90-day non-transplantation mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No